CLINICAL TRIAL: NCT02299128
Title: A Feasibility Study for a Randomized Controlled Trial on the Effectiveness of Early Physical Therapy Intervention for Patients With Dizziness After a Sports-Related Concussion
Brief Title: Effectiveness of Early Physical Therapy Intervention for Patients With Dizziness After a Sports-Related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walsh University (Other)
Collaborators: Children's Hospital Medical Center of Akron (Unknown); Kent State University (Other); American Academy of Orthopaedic Manual Physical Therapists (Other); Ohio Physical Therapy Association (Unknown)
Responsible Party: Principal Investigator, Jennifer Reneker, Assistant Professor, Walsh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-20
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Brain Concussion; Dizziness
MeSH Terms: conditions — Brain Concussion; Dizziness | interventions — Physical Therapy Modalities; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimally Therapeutic Treatment (Sham Comparator): Non-differential, prescriptive protocol of physical therapy treatment with minimal to no therapeutic benefit.
  Interventions: Other: Physical Therapy Treatment
- Skilled Treatment (Experimental): Differential treatment based on the results from the assessment. Physical Therapy treatment in this arm will be pragmatically designed and modified by the treating therapist. Treatments will include manual therapy to the cervical spine, neuromotor retraining (position sense and movement sense), habituation and adaptation exercises.
  Interventions: Other: Physical Therapy Treatment

INTERVENTIONS:
Other: Physical Therapy Treatment
  Other Names: Vestibular rehabilitation; Manual Therapy; Neuromotor training

SUMMARY:
Therefore, the purpose of this pilot study is to determine the feasibility of conducting a randomized clinical trial (RCT) on physical therapist treatment for dizziness after sports-related concussion. The specific research question for this pilot RCT is: What is the feasibility of conducting a RCT on athletes who have dizziness 10 or greater days after a sports-related concussion to explore the effectiveness of directed vestibular rehabilitation, neuromotor retraining, and/or manual physical therapy (PT) when compared to sham treatment? The findings of this study (for both feasibility and effect size) will be used to inform and direct revisions to the methods for a larger RCT on this population.

Primary Aims:

Specific Aim 1: Assess the feasibility of the following: recruitment and retention of participants, required resources for project management, and assessment of patient safety.

Specific Aim 2: Estimate the size of the effect between skilled physical therapist intervention and a sham treatment for the recovery rate for athletes with a concussion who have dizziness 10 - 14 days post-concussion.

DETAILED DESCRIPTION:
Study design: This study will be a pilot feasibility study of a RCT, randomized at the individual level.

Subjects:

The population of interest includes athletes who are seen by the physicians from a Sports Medicine Center (on site at Akron Children's Hospital (ACH) or at proxy locations, e.g. Walsh University or North Canton Children's Hospital Clinic) with a sports-related concussion. The specific population of interest is concussed patients who present for a medical assessment with dizziness as measured by the Post-Concussion Symptom Scale (PCS).

Sample Size and Sampling: Because this is a pilot study exploring the feasibility of the recruitment, retention and methods for a larger RCT, the sample is not intended to power a full scale study. It is standard for a pilot study to include at least 12 participants per arm of the study, however, because of the potential for loss to follow up the investigators plan to enroll 20 subjects per treatment group.

Study Subject Selection and Definitions: All patients who present to a Sports Medicine Center after an acute concussion (defined as any time between the event causing the concussion and up to 14 days after concussion) will complete the PCS. Within this 22 item scale, 7 items specify physical symptoms as components of the migraine cluster. These symptoms include: headaches, visual problems, dizziness, noise-light sensitivity, nausea/vomiting, balance problems, numbness/tingling. Although dizziness is the primary patient complaint being targeted, these other symptoms within the migraine cluster may also be present in addition to dizziness and may implicate a cervical, proprioceptive, and/or vestibular injury. For this reason, patients who report symptoms in the migraine cluster with one of the following criteria will be asked to enroll in the study at the initial assessment:

1. An initial score of at least 3 on the 7 point Likert scale for dizziness as a singular symptom OR
2. A score of 10 across the 7 items within the migraine cluster including a complaint of dizziness with at a score of at least 1 on the 7 point Likert scale OR
3. If findings from the objective assessment conducted by the physician indicate that postural/vestibular/ocular perception is abnormal.

Methods Allocation: At day10 after concussion, patients who enrolled in the study at their initial medical visit will be contacted by e-mail through Qualtrics and will be asked to complete the PCS a second time (if the patient sees the medical provider from Sports Medicine between day 10 and day 14, this will done on that same day). If at day 10 - 14 after the concussion was sustained, the patient continues to report dizziness with a score of at least 3 or a total score in the migraine cluster of at least 10 (including a score of at least 1 for dizziness) he/she will be randomized into one of the treatment groups using a random allocation sequence generator. If the patient does not meet the threshold of symptoms at day 10 - 14, they will receive standard medical care from the Sports Medicine physicians but will not be randomized into one of the PT treatment arms. One study investigator will be responsible for assignment into the treatment groups using a 1:1 allocation ratio.

Blinding: This study will be conducted as a double-blind trial whereby the physicians in the sports-medicine center, the patient participants, and their families will be blinded to the treatment allocation (sham or skilled) of patients throughout the study time. Blinding here is important to limit study bias because the physicians will determine one key outcome, the timeframe for return to play, and the athletes will report on the second key outcome, symptom severity on the PCS. The PTs performing the assessment and treatments will not be blinded to the allocation of the patients as they will be delivering the intervention. The same therapists will deliver both treatments (sham and skilled) based on allocation. Because the PTs cannot be blinded to the allocation of treatment, they will not determine the timeframe for return to play.

Patient follow-up: All patients allocated into one of the treatment arms will be followed for 4 consecutive weeks or until they are released for return to play by the sports medicine physician. All patients will continue to be followed by physicians in the sports medicine practice (as that is the standard of care).

Patient safety: Because this study is challenging the rest paradigm and using a progressive and active treatment to manage acute dizziness, it is not without risk. Patients will be carefully monitored during each visit to determine their response to treatment. Since the sham treatment incorporates no actual therapeutic activities, an exacerbation in symptoms is not expected. The skilled treatment group is pragmatic, allowing the treating therapists to determine the type and aggressiveness of each treatment session. This gives therapists the ability to modify the activity using their expert clinical judgment. For all subjects in the study, patient response between PT sessions will be monitored at the beginning of each PT treatment. If patient symptoms increase between therapy sessions, greater than the standard error of measure 6.3 points, treatment will be ceased and patients will be referred back to Sports Medicine for follow up. All adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 10 - 23 who have sustained a sports-related concussion.
* Sports will include participation in any organized sporting activity (including club teams, recreational sports, or school teams).
* Patients with a history of learning disorders, use of medication (including psychotropics or narcotics) will be included.

Exclusion Criteria:

* Patients younger than 10 years or older than 23 years of age.
* If the patient has a concussion that was sustained during activities other than sports-related (bicycle accident, motor vehicle accident, or other non-sports related activities) they will not be enrolled in this study.
* Athletes with concussion who have symptoms but none of their complaints include dizziness or indicate a postural/vestibular/ocular or perceptual abnormality will be excluded.
* Finally, athletes who present to the sports-medicine physician for an initial assessment greater than 14 days after they sustained a concussion will be excluded.

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Symptom recovery as measured by the Post Concussion Symptom (PCS) Score | Final visit (by the end of 4 weeks of treatment)
  7 point Likert scale (0 - 6) rating the severity of 22 symptoms commonly associated with concussion.
Return to Play (RTP) | Final visit (by the end of 4 weeks of treatment)
  Five stage progressive increase in physical activity ranging from minimal exertion to full contact in a game

SECONDARY OUTCOMES:
Change Score of Functional Gait Assessment | Initial assessment and final visit (by the end of 4 weeks of treatment)
  Used to test balance with gait activities.
Change score of Vertigo Symptom Scale - Short Form | Initial assessment and final visit (by the end of 4 weeks of treatment)
  Frequency of various types and durations of sensation of dizziness
Global Response to Treatment | Final Visit (by the end of 4 weeks of treatment)
  Global perception of change in physical symptoms from the beginning of treatment to the end

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Reneker, MSPT, Principal Investigator — Walsh University
Locations (1):
- Walsh University, North Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No